CLINICAL TRIAL: NCT01626092
Title: Treatment of High Risk, Inherited Lysosomal and Peroxisomal Disorders by Reduced-Intensity Hematopoietic Cell Transplantation and Low-Dose Total Body Irradiation With Marrow Boosting by Volumetric-Modulated Arc Therapy (VMAT)
Brief Title: Reduced-Intensity Hematopoietic Stem Cell Transplant for High Risk Lysosomal and Peroxisomal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS147; MT2011-24 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Lysosomal Storage Disease; Peroxisomal Disorder
Keywords: bone marrow transplantation; reduced intensity conditioning; Adrenoleukodystrophy; Metachromatic Leukodystrophy; Globoid Cell Leukodystrophy; Wolman's disease; GM1 gangliosidosis; Tay Sachs disease; Sanfilippo syndrome; Sandhoff disease; inherited metabolic; I-cell disease; mucolipidosis II
MeSH Terms: conditions — Lysosomal Storage Diseases; Peroxisomal Disorders; Adrenoleukodystrophy; Leukodystrophy, Metachromatic; Leukodystrophy, Globoid Cell; Wolman Disease; Gangliosidosis, GM1; Tay-Sachs Disease; Mucopolysaccharidosis III; Sandhoff Disease; Mucolipidoses | interventions — Alemtuzumab; Clofarabine; Melphalan; Whole-Body Irradiation; Radiotherapy, Intensity-Modulated; Hematopoietic Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-To-Treat Patients (Experimental): Patients with high-risk lysosomal and peroxisomal disorders treated with preparative regimen (Campath-1H 0.3 mg/kg intravenous (IV) on days -12 through -8, clofarabine 40 mg/m^2 IV on days -9 through -5, melphalan 140 mg/m^2 IV on day -4 and Total Body Irradiation with Marrow Boosting [ first dose of 200 cGy single dose; 5 doses of 160cGy for marrow boosting - 1000cGy cumulative exposure] by Volumetric-Modulated Arc Therapy [VMAT] on days -3 through -1). Hematopoietic stem cell transplantation will be infused on Day 0. Post-transplant immunosuppression to follow: Mycophenolate mofetil (MMF) begin day -3 and continue to day +30 or 7 days after engraftment, whichever is later; Cyclosporine A (CsA) begin day -3 and then taper at day +100 if related donor, day +180 for unrelated donor.
  Interventions: Drug: Campath-1H; Drug: Clofarabine; Drug: Melphalan; Radiation: Total Body Irradiation with Marrow Boosting; Biological: Hematopoietic stem cell transplantation; Drug: Cyclosporine A; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Campath-1H — A daily dose of 0.3 mg/kg IV over 2 hours will be administered on days - 12, -11, -10, -9, and -8.
  Other Names: alemtuzumab-1H
Drug: Clofarabine — A daily dose of 40 mg/m2 will be administered IV over 2 hours on days -9,
  -8, -7, -6, and -5.
  Other Names: Clolar
Drug: Melphalan — A single dose of 140 mg/m2 will be given IV on day -4 over 15 minutes.
  Other Names: Alkeran
Radiation: Total Body Irradiation with Marrow Boosting — 1. Dose to total body 200 cGy in single dose
  2. Dose to bone marrow of the following bones 800 cGy in 5 divided daily fractions (160 cGy x 5 doses ). Treated with up to 3 abutting VMAT photon arcs from top of head to maximum inferior border.
  Other Names: Volumetric-Modulated Arc Therapy (VMAT)
Biological: Hematopoietic stem cell transplantation — Patients will be transplanted using either a related or unrelated allograft. The cell source may be marrow, peripheral blood or cord blood based on donor availability.
Drug: Cyclosporine A — Patients will receive CsA therapy beginning on day -3. Dosing of CsA will be 2.5 mg/kg/dose IV; if the recipient body weight is <40 kg, dosing will be 3 times daily, and if > 40 kg, twice daily. An attempt will be made to maintain a trough cyclosporine level of 200 mg/L to 400 mg/L.
  Other Names: CsA
Drug: Mycophenolate mofetil — Patients will receive mycophenolate mofetil (MMF) therapy beginning on day -3. Dosing of MMF will be 1 gram three times daily (total daily dose 3 grams/day) if the recipient is >50 kg, or 15 mg/kg/dose three times daily if the recipient is ≤50 kg. The same dosage is used orally or intravenously.
  Other Names: MMF

SUMMARY:
This study is designed to test the ability to achieve donor hematopoietic engraftment while maintaining low rates of transplant-related mortality (TRM) in patients with high-risk lysosomal and peroxisomal disorders using a novel conditioning regimen for hematopoietic cell transplantation (HCT). After a reduced-intensity conditioning regimen using volumetric-modulated arc therapy (VMAT)-delivered low-dose total body irradiation (TBI) with highly conformal marrow boosting, patients will be transplanted using either a related or unrelated allograft. The cell source may be marrow, peripheral blood or cord blood based on donor availability.

DETAILED DESCRIPTION:
The conditioning regimen consists of alemtuzumab (Campath-1H), clofarabine, melphalan, and VMAT-delivered low-dose TBI with boosted marrow irradiation. Additional graft-versus-host disease prophylaxis consists of mycophenolate mofetil and cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Adrenoleukodystrophy (ALD): Patients from 0-55 years of age diagnosed with ALD as determined by very long chain fatty acid testing will be eligible for this protocol if they have evidence of cerebral or cerebellar disease based on MRI testing,
* Metachromatic Leukodystrophy (MLD): Patients from 0-55 years of age diagnosed with MLD as determined by arylsulfatase A activity.
* Globoid Cell Leukodystrophy (GLD): Patients from 0-55 years of age diagnosed with GLD as determined by galactocerebrosidase activity will be eligible for this protocol
* Wolman's disease, GM1 gangliosidosis, Tay Sachs disease, Sanfilippo syndrome, Sandhoff disease or other inherited metabolic diseases including but not limited to I-cell disease (mucolipidosis II): Patients who are determined to be sufficiently advanced or high risk based on the following reasons:

  * Symptomatic disease, as based on neurologic examination or evidence of deterioration based on subsequent neuropsychologic evaluations.
  * Evidence of an expected poor outcome based on genetic testing or a prior family history of aggressive disease.
  * Other metabolic disorders, including but not limited to I-cell disease, that are deemed to be high-risk for a poor outcome with a standard transplant regimen due to anticipated toxicity based on experience gained at the University of Minnesota or other centers.
* Donor Availability

  * Transplantation using sufficiently matched related donors (such as matched siblings) or unrelated donors will be considered. Both granulocyte-colony stimulating factor (G-CSF) stimulated peripheral blood grafts and bone marrow grafts will be considered, although bone marrow will be the priority.
  * Cord blood grafts, both related and unrelated, are also eligible. As this protocol will use a reduced intensity regimen, this protocol will use the current recommendations of the University of Minnesota for choosing cord blood grafts. If a single cord blood unit cell dose is insufficient, double cord transplantation should be considered if sufficiently matched cord blood units are available. The priority of choosing cord blood donors is based on the current institutional recommendations.
  * Exclusion of Metabolic Disorder Carrier Status from related donor and unrelated cord blood grafts as appropriate for primary disease.
* Adequate Organ Function - Measured within 30 days of study enrollment
* Signed consent

Exclusion Criteria:

* Inability to receive total body irradiation (TBI) with marrow boosting per protocol guidelines as determined by the Radiation Oncologist
* Pregnant - Menstruating females must have a negative serum pregnancy test within 14 days of treatment start.
* Advanced Disease Exclusion: Following evaluation, if a consensus of the members of the Inherited Metabolic and Storage Disease Program is that a patient is too advanced to benefit in a measurable and meaningful way from transplant, this will be communicated to the family, and transplant will not be offered.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weston Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent-To-Treat Patients: Patients with high-risk lysosomal and peroxisomal disorders treated with preparative regimen (Campath-1H 0.3 mg/kg intravenous (IV) on days -12 through -8, clofarabine 40 mg/m^2 IV on days -9 through -5, melphalan 140 mg/m^2 IV on day -4 and Total Body Irradiation with Marrow Boosting [ first dose of 200 cGy single dose; 5 doses of 160cGy for marrow boosting - 1000cGy cumulative exposure] by Volumetric-Modulated Arc Therapy [VMAT] on days -3 through -1). Hematopoietic stem cell transplantation will be infused on Day 0. Post-transplant immunosuppression to follow: Mycophenolate mofetil (MMF) begin day -3 and continue to day +30 or 7 days after engraftment, whichever is later; Cyclosporine A (CsA) begin day -3 and then taper at day +100 if related donor, day +180 for unrelated donor.
  Campath-1H: A daily dose of 0.3 mg/kg IV over 2 hours will be administered on days - 12, -11, -10, -9, and -8.
  Clofarabine: A daily dose of 40 mg/m2 will be administered IV over 2 hours on days -9,
Period: Overall Study
Arm/Group | Intent-To-Treat Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intent-To-Treat Patients: Patients with high-risk lysosomal and peroxisomal disorders treated with preparative regimen (Campath-1H 0.3 mg/kg intravenous (IV) on days -12 through -8, clofarabine 40 mg/m^2 IV on days -9 through -5, melphalan 140 mg/m^2 IV on day -4 and Total Body Irradiation with Marrow Boosting [ first dose of 200 cGy single dose; 5 doses of 160cGy for marrow boosting - 1000cGy cumulative exposure] by Volumetric-Modulated Arc Therapy [VMAT] on days -3 through -1). Hematopoietic stem cell transplantation will be infused on Day 0. Post-transplant immunosuppression to follow: Mycophenolate mofetil (MMF) begin day -3 and continue to day +30 or 7 days after engraftment, whichever is later; Cyclosporine A (CsA) begin day -3 and then taper at day +100 if related donor, day +180 for unrelated donor.
  Campath-1H: A daily dose of 0.3 mg/kg IV over 2 hours will be administered on days - 12, -11, -10, -9, and -8
  Clofarabine: A daily dose of 40 mg/m2 will be administered IV over 2 hours on days -9
Arm/Group | Intent-To-Treat Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Donor (Allogeneic) Hematopoietic Engraftment
Description: Number of patients who achieve hematopoietic engraftment - assessment of nucleated peripheral blood cells for donor (allogeneic) chimerism following this reduced-intensity HCT.
Time Frame: Day 100 Following Hematopoietic Cell Transplant (HCT)
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat Patients
Number analyzed (Participants) | 3
participants | 1

2. Secondary Outcome: Transplant-Related Mortality
Description: Incidence of death due to complications of HCT following this reduced-intensity conditioning regimen.
Time Frame: Day 100 following HCT
Measure: Number; unit: participants
Arm/Group | Intent-To-Treat Patients
Number analyzed (Participants) | 3
participants | 0

3. Secondary Outcome: Neurologic Outcomes
Description: Depending upon underlying primary disease, a combination of evaluative tools (e.g. brain magnetic resonance imaging (MRI), clinical neurologic exam, neuropsychologic testing, electromyography) will be applied for assessment of neurologic function and how it may be affected by this reduced-intensity HCT regimen.
Time Frame: Changes from Baseline, Days 30, 60, 100, Year 1, Year 2, Year 3 Following HCT
Population: None of the 3 patients enrolled in the study were evaluable for this outcome. Two had a repeat transplant and one was lost to follow-up.
Arm/Group | Intent-To-Treat Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intent-To-Treat Patients
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intent-To-Treat Patients (N=3)
Hearing loss (Ear and labyrinth disorders) | 1
Decreased vision (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 3
Acid reflux (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Positive blood culture - Staphylococcus aureus (Infections and infestations) | 1
Positive blood culture - Escherichia coli (Infections and infestations) | 1
Fever (Infections and infestations) | 1
BK viruria (Infections and infestations) | 1
Adenoviremia (Infections and infestations) | 1
Acute radiation syndrome (Injury, poisoning and procedural complications) | 1
Graft failure (Injury, poisoning and procedural complications) | 3
Elevated lipase (Investigations) | 1
Serum amylase increased (Investigations) | 2
Hypogammaglobulinemia (Investigations) | 1
Elevated ALT (Investigations) | 1
Elevated AST (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 1
Muscle spasms (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Decreased oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes